CLINICAL TRIAL: NCT05467072
Title: Post-Marketing Clinical Follow-up of an Annular Closure System
Brief Title: PMCFU of an Annular Closure System
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Intrinsic Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: CP-013
Record Dates: First submitted 2022-07-18; First posted 2022-07-20 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Lumbar Disc Herniation
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Discectomy + annular closure: All patients treated with lumbar discectomy and implantation of an annular closure device
  Interventions: Device: Annular closure

INTERVENTIONS:
Device: Annular closure — Lumbar discectomy patients treated with Annular Closure Device BARRICAID

SUMMARY:
The purpose of this retrospective chart review study is to collect the data that will be used to provide clinical evidence to support the post-market surveillance program.

DETAILED DESCRIPTION:
Retrospective chart review of patients treated with lumbar discectomy and annular closure. Review of patient charts through 3 month post op, for analysis of symptomatic lumbar reherniation at the index level.

ELIGIBILITY:
Inclusion Criteria:

* Records for any subject treated with a Barricaid annular closure device will be considered for inclusion into the study

Exclusion Criteria:

* Records for any subject treated without a Barricaid annular closure device will be considered for exclusion

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient previously treated with lumbar discectomy and annular closure, with 3 month post op follow up data available
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-09-27 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Symptomatic reherniation | 3 months post op
  Reherniation of the index lumbar disc level, with patient symptoms (back or leg pain)

CONTACTS AND LOCATIONS:
Overall Officials: David H Kim, MD, Study Chair — New England Baptist Hospital
Locations (1):
- Orthopedic Institute of Western Kentucy, Paducah, Kentucky, United States